CLINICAL TRIAL: NCT07001514
Title: The Effect of Evening Technology Use With Calming vs. Exciting Content on Sleep Architecture in Older Adults: A Crossover Randomized Controlled Trial
Brief Title: Evening Screen Content and Sleep Architecture in Older Adults: Crossover RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blekinge Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: BTH-6.1.1-0093-2025
Record Dates: First submitted 2025-05-12; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calming Digital Content (Experimental): Participants will watch calming digital content - specifically, nature documentaries narrated by Sir David Attenborough - for 30 to 60 minutes within one hour before bedtime. Sleep outcomes will be assessed using EEG recordings and subjective sleep quality logs.
  Interventions: Behavioral: Calming digital content
- Exciting Digital Content (Experimental): Participants will engage with exciting digital content by playing the word-based game Ruzzle for 30 to 60 minutes within one hour before bedtime. Sleep outcomes will be evaluated using EEG measurements and subjective sleep assessments.
  Interventions: Behavioral: Exciting Digital Content
- Non-Digital Pre-Sleep Activity (Active Comparator): Participants will engage in a non-digital activity by reading a physical, non-fiction book of their choice for 30 to 60 minutes within one hour before bedtime. No digital screens will be used. Sleep outcomes will be monitored via EEG data and self-reported sleep quality measures.
  Interventions: Behavioral: Non-digital book reading

INTERVENTIONS:
Behavioral: Calming digital content — Participants watch a curated selection of soothing documentaries narrated by Sir David Attenborough for 30-60 minutes each evening during one hour before bedtime.
  Other Names: digital; nature documentary
  Arms: Calming Digital Content
Behavioral: Exciting Digital Content — Participants engage with the interactive word-based game Ruzzle for 30-60 minutes each evening during one hour before bedtime, designed to provide mental stimulation.
  Other Names: Digital; Ruzzle; Game
  Arms: Exciting Digital Content
Behavioral: Non-digital book reading — Participants read a non-fiction book of their choice for the same duration, avoiding all digital screens during one hour before bedtime before bedtime.
  Other Names: book reading
  Arms: Non-Digital Pre-Sleep Activity

SUMMARY:
Title

The Effect of Evening Technology Use with Calming vs. Exciting Content on Sleep Architecture in Older Adults: A Crossover Randomized Controlled Trial

Background

The study explores how evening use of digital devices with different types of content (calming vs. exciting) affects sleep in older adults. While technology's effects on sleep have been studied in younger populations, its specific impacts on older adults remain under-researched. This study fills that gap by focusing on subjective and objective sleep measures.

Objectives and Research Questions

Objective: Compare the effects of calming digital content, exciting digital content, and non-digital activities on sleep architecture.

Key Questions:

How does content type impact sleep architecture and quality? Does calming content lead to better sleep outcomes than exciting content? Are there subjective differences in sleep quality across conditions?

DETAILED DESCRIPTION:
This study will compare the effects of watching calming (nature documentaries), playing exciting digital games like Ruzzle, and reading a physical book on older adults' subjective and objective sleep quality. This will be a randomized crossover trial. The investigators will exclude participants with diagnosed sleep disorders, Severe cognitive impairment, Use of sleep-affecting medications such as melatonin or benzodiazepines, or Irregular sleep schedules. A sample size of approximately 50 participants (49-51) will be recruited.

All the participants will have all three intervention periods with washout periods in between. During every intervention week, participants will fill out a quick nightly log about their sleep and what tech they used (smartphone, tablet, or a laptop/computer). During sleep, they will wear a comfy EEG headband measuring their sleep stages.

Because everyone eventually does all three conditions, the investigators can compare each person's own results and get more precise answers with fewer people.

The investigators will analyze the data and perform a statistical analysis. The study will be reported in the manuscript and published in a reputable journal.

ELIGIBILITY:
Inclusion Criteria

1. Age 60 - 75 years
2. Regular evening use of digital devices (e.g., smartphones or tablets)
3. Willing and able to wear an EEG headband for sleep monitoring throughout the intervention

Exclusion Criteria:

1. Diagnosed sleep disorder
2. Severe cognitive impairment
3. Current use of medications that significantly influence sleep (e.g., melatonin, benzodiazepines)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sleep architecture REM | Nightly during each participant's 7-day intervention periods - Week 1 (Days 1-7), Week 3 (Days 15-21), and Week 5 (Days 29-35) after that participant's enrollment; up to 5 weeks per participant.
  Sleep architecture containing sleep stages REM - Random eye movement stage.
Sleep architecture Deep Sleep | Nightly during each participant's 7-day intervention periods - Week 1 (Days 1-7), Week 3 (Days 15-21), and Week 5 (Days 29-35) after that participant's enrollment; up to 5 weeks per participant.
  Sleep architecture containing sleep stages, Deep sleep
Sleep architecture, light sleep | Nightly during each participant's 7-day intervention periods - Week 1 (Days 1-7), Week 3 (Days 15-21), and Week 5 (Days 29-35) after that participant's enrollment; up to 5 weeks per participant.
  Sleep architecture containing sleep stages, light sleep
Sleep latency (time to fall asleep) | Nightly during each participant's 7-day intervention periods - Week 1 (Days 1-7), Week 3 (Days 15-21), and Week 5 (Days 29-35) after that participant's enrollment; up to 5 weeks per participant.
  time to fall asleep- through EEG headband
Total sleep time (TST) | Nightly during each participant's 7-day intervention periods - Week 1 (Days 1-7), Week 3 (Days 15-21), and Week 5 (Days 29-35) after that participant's enrollment; up to 5 weeks per participant.
  Total amount or duration of sleep
Sleep efficiency (SE) | Nightly during each participant's 7-day intervention periods - Week 1 (Days 1-7), Week 3 (Days 15-21), and Week 5 (Days 29-35) after that participant's enrollment; up to 5 weeks per participant.
  Sleep efficiency (SE)- Sleep efficiency is the percentage of time in bed actually spent sleeping. It is calculated by dividing total sleep time by total time spent in bed and multiplying by 100. Higher sleep efficiency suggests less wakefulness during the night and better overall sleep quality.
Wake up after sleep onset (WASO). | Nightly during each participant's 7-day intervention periods - Week 1 (Days 1-7), Week 3 (Days 15-21), and Week 5 (Days 29-35) after that participant's enrollment; up to 5 weeks per participant.
  Wake up after sleep onset (WASO).WASO measures the cumulative amount of time a participant spends awake after initially falling asleep, until final morning awakening. Elevated WASO values may indicate fragmented or disrupted sleep, which can negatively affect sleep quality and daytime functioning.

SECONDARY OUTCOMES:
Subjective sleep quality | Each morning from Day 1 through Day 35 after each participant's enrollment, covering all intervention and washout weeks; up to 5 weeks per participant
  Single-Item Sleep Quality Scale. Range 0 (Terrible) to 10 (Excellent)
Comfort of using the EEG headband | Each morning during each participant's 7-day intervention periods - Week 1 (Days 1-7), Week 3 (Days 15-21), and Week 5 (Days 29-35) after that participant's enrollment; up to 5 weeks per participant
  How comfortable do you find wearing the EEG headband at night?
  1. - Very uncomfortable
  2. - Slightly uncomfortable
  3. - Neither comfortable nor uncomfortable
  4. - Somewhat comfortable
  5. - Very comfortable
Intervention Adherence | Each morning during each participant's 7-day intervention periods - Week 1 (Days 1-7), Week 3 (Days 15-21), and Week 5 (Days 29-35) after that participant's enrollment; up to 5 weeks per participant
  Participants will be asked whether they were able to complete the assigned evening activity the previous night. If the answer is "yes," they will also report how long they engaged in the intervention (in minutes). This self-report measure will help evaluate the feasibility and real-world compliance with each intervention condition.

OTHER OUTCOMES:
Baseline survey | Baseline (Day 0, at enrollment; one-time survey)
  Before the first intervention phase, participants complete a baseline survey assessing:
  Sociodemographic characteristics (Gender, Living status, economic situation, working status, how many hours do you work, education status).
  Subjective sleep health (SATED 3 item likert scale instrument with five questions).
  Sleeping habits (sleep medication use?, Sleep-schedule regularity,Daytime napping, Evening screen exposure, Sleep disruption by physical symptoms (pain,itching), Sleep disruption by psychological factors, Night-time technology use, Nocturia).
  Chronotype (The reduced Morningness-Eveningness Questionnaire), general health status (0 bad to 4 excellent).
  Technology use (On average, how often have you used the INTERNET on your computer, tablet and smartphone in the last three months?).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Anderberg, PhD, Principal Investigator — Blekinge Institute of Technology
Locations (1):
- Blekinge Institute of Technology, Karlskrona, Blekinge County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared publicly because the study involves sensitive sleep and health-related data from older adult participants. To protect participant privacy and confidentiality, the data will remain anonymized and securely stored for analysis by the research team only. Public sharing of individual-level data is not planned.